CLINICAL TRIAL: NCT00512707
Title: Androgen Modulation of Response to Selective Phosphodiesterase Inhibitors in Erectile Dysfunction
Brief Title: Effect of Testosterone in Men With Erectile Dysfunction
Acronym: TED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-25065; R01HD047722-01A1 (NIH)
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Erectile Dysfunction; Testosterone Deficiency; Diabetes
Keywords: testosterone; erectile dysfunction; sildenafil
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus | interventions — Sildenafil Citrate; Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Testosterone Gel (Experimental): Active Testosterone Gel and on demand use of sildenafil citrate (3 tablets per week). Starting dose of 50 mg. Titrated to 100 mg or 25 mg depending on efficacy and tolerability. Begins as open label run in period for 3 - 6 weeks, and continues during the placebo-controlled testosterone gel intervention for 16 weeks.
  Interventions: Drug: Sildenafil citrate (open label); Drug: Testosterone gel
- Placebo Gel (Placebo Comparator): Placebo Gel and on demand use of sildenafil citrate (3 tablets per week). Starting dose of 50 mg. Titrated to 100 mg or 25 mg depending on efficacy and tolerability. Begins as open label run in period for 3 - 6 weeks, and continues during the placebo-controlled testosterone gel intervention for 16 weeks.
  Interventions: Drug: Sildenafil citrate (open label); Other: Placebo gel

INTERVENTIONS:
Drug: Sildenafil citrate (open label) — On demand use of sildenafil citrate (3 tablets per week). Starting dose of 50 mg. Titrated to 100 mg or 25 mg depending on efficacy and tolerability. Begins as open label run in period for 3 - 6 weeks, and continues during the placebo-controlled testosterone gel intervention for 16 weeks.
  Other Names: Viagra (Pfizer Inc.)
Drug: Testosterone gel — Testosterone Gel 1%: Starting active dose 10 g/day. Increased to 15 g/day or decreased to 5 g/day in order to attain morning total testosterone level between 500 - 1000 ng/dL. Blinding achieved by combining a total of 3 tubes of active or placebo gel, applied to upper arms and shoulders each day.
  Other Names: Testim (Auxilium Pharmaceuticals, Inc.)
  Arms: Active Testosterone Gel
Other: Placebo gel — 3 tubes of placebo gel equivalent to the amount of the testosterone gel will be applied during the placebo-controlled testosterone gel intervention for 16 weeks..
  Arms: Placebo Gel

SUMMARY:
The purpose of this placebo-controlled study is to determine if testosterone replacement therapy, administered by transdermal gel, can improve the response to sildenafil (Viagra R) treatment in men who have erectile dysfunction (ED) and low testosterone levels.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, parallel-group, randomized clinical trial in men, 40-70 years of age, who present with mild to moderate erectile dysfunction and have androgen deficiency defined as serum total testosterone level below 300 ng/dL, measured by liquid chromatography tandem mass spectrometry, LC-MS/MS (15) and/or free testosterone level (measured by equilibrium dialysis) below 50 pg/ml. Sexual function assessments will include validated erectile function questionnaires (IIEF), sexual activity diaries, sexual desire, partner interaction and intimacy, affects balance scale, mood, ED-related quality of life, and penile rigidity in response to a visual erotic stimulus. The initial assessment will be made prior to treatment with sildenafil citrate, i.e., in subjects who are naïve to or withdrawn from PDE5 inhibitors and/or testosterone. Participants will then be allotted three sildenafil citrate tablets per week (12 pills per month), but will not use more than one tablet within any 24-hour period. During the Sildenafil-Dose Optimization period, subjects naïve to sildenafil citrate will start with a 50 mg dose. Those who have used sildenafil citrate in the past will take the same dose that was found to be efficacious for them. After three weeks, the dose of sildenafil citrate will be increased to 100-mg in non-responders. For those who cannot tolerate the 50-mg dose, a dose of 25 mg will be given. After three weeks on the optimized dose of sildenafil citrate, subjects will undergo a second evaluation of sexual function. They will then be randomly assigned to receive this optimized dose of sildenafil citrate with either placebo gel (15 g per day) or active testosterone gel (10 g active gel + 5 g placebo gel per day). The daily dose of active testosterone gel was selected to increase average serum into the upper-half of the normal range for healthy, young men (e.g., 500-1000 ng/dL). In order to assure that serum testosterone levels are in the target range (500-1000 ng/dL), testosterone dose will be adjusted by an unblinded individual two to three weeks after initiation of testosterone/placebo treatment, based on the measurement of serum testosterone levels. If the average testosterone level is less than 500 ng/dL, the daily dose will be increased to 15g of active gel. If the average testosterone is greater than 1,000 ng/dL, the daily dose will be decreased to 5 g of active gel (and 10 g of placebo gel). This dose adjustment will take effect at week 4 (day 28) of treatment. Subjects will be treated for an additional 12-weeks with sildenafil citrate and the optimized dose of testosterone gel or placebo gel. Sexual function will be evaluated at the end of this treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Men, 40-70 years of age, in a stable relationship, with mild to moderate erectile dysfunction for at least 6 months; defined as an IIEF-EF domain score between 11 and 25 (mild to moderate ED)
* Neutral or extremely dissatisfied with one's sex life
* Presence of androgen deficiency defined as serum total testosterone level less than 300 ng/dL (measured by LC-MS/MS) and/or free testosterone level (measured by equilibrium dialysis) less than 50 pg/ml.
* Able to understand the nature of the study and provide written, informed consent

Exclusion Criteria:

* Contraindication for use of testosterone, e.g., history of prostate or breast cancer
* benign prostatic hyperplasia with AUA/IPSS symptom scores of 21 or greater
* erythrocytosis (hematocrit >50% at baseline)
* untreated, severe sleep apnea
* serum PSA levels >4 ug/L will be excluded unless they have had a urologic evaluation in the past three months to exclude prostate cancer.
* Contraindication for use of sildenafil, e.g., symptomatic coronary artery disease taking long-acting or short-acting nitrate drugs on a regular basis.
* Symptomatic postural hypotension
* Congestive heart failure with class III or IV symptoms
* History of myocardial infarction or stroke within the past six months
* Primary diagnosis of another sexual disorder such as premature ejaculation
* AST, ALT, alkaline phosphatase elevation greater than three times the upper limit of normal, creatinine greater than 2 mg/dL.
* Currently taking testosterone or oral androgen precursors; unless willing to discontinue their use for 4 weeks (oral precursors or transdermal testosterone patch or gel) or 6 weeks (if injectable testosterone) before the initial screen visit.
* Currently taking medications that affect androgen metabolism, action, or clearance (dilantin, phenobarbital, aldactone, flutamide, finasteride).
* Uncontrolled diabetes mellitus or diabetes mellitus, e.g., if their baseline hemoglobin A1C is less than 8.5%.
* Structural abnormalities of the penis, including Peyronie's disease, will be excluded.
* Men who are taking medications for erectile dysfunction, including sildenafil, must stop using these medications for at least 4 weeks before starting Visit 2.
* DSM-IV criteria for an Axis I psychiatric disorder within the past year, including depression; use of psychotropic medication for at least six months, or dementia is also an exclusion.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee H, Hwang EC, Oh CK, Lee S, Yu HS, Lim JS, Kim HW, Walsh T, Kim MH, Jung JH, Dahm P. Testosterone replacement in men with sexual dysfunction. Cochrane Database Syst Rev. 2024 Jan 15;1(1):CD013071. doi: 10.1002/14651858.CD013071.pub2. PMID 38224135
- [Derived] Wilson E, Gannon H, Chimhini G, Fitzgerald F, Khan N, Lorencatto F, Kesler E, Nkhoma D, Chiyaka T, Haghparast-Bidgoli H, Lakhanpaul M, Cortina Borja M, Stevenson AG, Crehan C, Sassoon Y, Hull-Bailey T, Curtis K, Chiume M, Chimhuya S, Heys M. Protocol for an intervention development and pilot implementation evaluation study of an e-health solution to improve newborn care quality and survival in two low-resource settings, Malawi and Zimbabwe: Neotree. BMJ Open. 2022 Jul 5;12(7):e056605. doi: 10.1136/bmjopen-2021-056605. PMID 35790332
- [Derived] Spitzer M, Bhasin S, Travison TG, Davda MN, Stroh H, Basaria S. Sildenafil increases serum testosterone levels by a direct action on the testes. Andrology. 2013 Nov;1(6):913-8. doi: 10.1111/j.2047-2927.2013.00131.x. Epub 2013 Sep 18. PMID 24106072
- [Derived] Spitzer M, Basaria S, Travison TG, Davda MN, DeRogatis L, Bhasin S. The effect of testosterone on mood and well-being in men with erectile dysfunction in a randomized, placebo-controlled trial. Andrology. 2013 May;1(3):475-82. doi: 10.1111/j.2047-2927.2013.00075.x. Epub 2013 Mar 15. PMID 23494931
- [Derived] Spitzer M, Basaria S, Travison TG, Davda MN, Paley A, Cohen B, Mazer NA, Knapp PE, Hanka S, Lakshman KM, Ulloor J, Zhang A, Orwoll K, Eder R, Collins L, Mohammed N, Rosen RC, DeRogatis L, Bhasin S. Effect of testosterone replacement on response to sildenafil citrate in men with erectile dysfunction: a parallel, randomized trial. Ann Intern Med. 2012 Nov 20;157(10):681-91. doi: 10.7326/0003-4819-157-10-201211200-00004. PMID 23165659

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone: Active Testosterone Gel
  Sildenafil citrate (open label): On demand use of sildenafil citrate (3 tablets per week). Starting dose of 50 mg. Titrated to 100 mg or 25 mg depending on efficacy and tolerability. Begins as open label run in period for 3 - 6 weeks, and continues during the placebo-controlled testosterone gel intervention for 16 weeks.
  Testosterone gel 1% (active or placebo): Testosterone Gel 1%: Starting active dose 10 g/day. Increased to 15 g/day or decreased to 5 g/day in order to attain morning total testosterone level between 500 - 1000 ng/dL. Blinding achieved by combining a total of 3 tubes of active or placebo gel, applied to upper arms and shoulders each day.
  Topical testosterone gel 1%: Testosterone Gel: Starting dose 10 g/day. Increased to 15 g/day or decreased to 5 g/day in order to attain morning total testosterone level between 500 - 1000 ng/dL. Blinded achieved by combining a total of 3 tubes of active or placebo gel.
- Placebo: Placebo Gel
  Sildenafil citrate (open label): On demand use of sildenafil citrate (3 tablets per week). Starting dose of 50 mg. Titrated to 100 mg or 25 mg depending on efficacy and tolerability. Begins as open label run in period for 3 - 6 weeks, and continues during the placebo-controlled testosterone gel intervention for 16 weeks.
  Testosterone gel 1% (active or placebo): Testosterone Gel 1%: Starting active dose 10 g/day. Increased to 15 g/day or decreased to 5 g/day in order to attain morning total testosterone level between 500 - 1000 ng/dL. Blinding achieved by combining a total of 3 tubes of active or placebo gel, applied to upper arms and shoulders each day.
Period: Overall Study
Arm/Group | Testosterone | Placebo
Started | 70 | 70
Completed | 60 | 58
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 5 | 11
Not completed — Developed skin irritation | 2 | 1
Not completed — Developed a hematocrit exceeding 0.54 | 2 | 0
Not completed — Unable to tolerate the smell of the gel | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristic are provided prior to sildenafil administration (week -7)
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (8.3) | 54.6 (8.5) | 54.9 (8.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 70 | 70 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Based on the number of participants who responded.
  Participants
    Race: number analyzed (Participants) | 68 | 70 | 138
    Race: Black | 28 | 33 | 61
    Race: White | 36 | 32 | 68
    Race: Other | 4 | 5 | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (6.4) | 32.7 (6.0) | 32.1 (6.2)
Diabetes mellitus [Count of Participants; unit: Participants] | 13 | 14 | 27
Hypertension [Count of Participants; unit: Participants] | 29 | 27 | 56
Cardiovascular disease [Count of Participants; unit: Participants] | 35 | 32 | 67
Total testosterone level [Mean (Standard Deviation); unit: ng/dL] | 248 (62) | 254 (68) | 251 (65)
Total testosterone level <250 ng/dL [Count of Participants; unit: Participants] | 31 | 28 | 59
Free testosterone level [Mean (Standard Deviation); unit: pg/mL] | 45 (15) | 47 (16) | 46 (15)
International Index of Erectile Function (IIEF) [Mean (Standard Deviation); unit: units on a scale] — IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
  units on a scale
    Erectile function | 12.2 (5.9) | 12.0 (6.5) | 12.1 (6.2)
    Orgasmic function | 5.1 (3.0) | 5.4 (3.1) | 5.3 (3.1)
    Sexual desire | 5.6 (1.9) | 5.6 (1.9) | 5.6 (1.9)
    Intercourse satisfaction | 6.1 (3.4) | 6.0 (3.6) | 6.0 (3.5)
    Overall satisfaction | 4.3 (1.9) | 4.5 (2.1) | 4.4 (2.0)
    Composite IIEF | 33 (13) | 33 (14) | 33 (13)
Sexual Encounter Profile (SEP) [Mean (Standard Deviation); unit: events/week] — Sexual Encounter Profile (SEP) diaries assesses frequency of sexual activity, sildenafil use, vaginal penetration, completion of intercourse with ejaculation, and overall satisfaction with sexual encounters. Minimum value is 0 with no maximum limit, wherein higher values representing better sexual encounter.
  events/week
    Sexual encounter attempts | 2.5 (1.4) | 2.3 (1.3) | 2.4 (1.3)
    Vaginal penetrations | 1.5 (1.3) | 1.4 (1.1) | 1.4 (1.2)
    Ejaculations | 0.92 (1.11) | 1.14 (1.15) | 1.02 (1.13)
    Overall satisfied with sexual encounters | 0.49 (0.71) | 1.07 (1.39) | 0.76 (1.12)
Successful sexual Intercourse in Sexual Encounter Profile (SEP) [Mean (Standard Deviation); unit: percentage of successful intercourse] — Sexual Encounter Profile (SEP) diaries assesses frequency of sexual activity, sildenafil use, vaginal penetration, completion of intercourse with ejaculation, and overall satisfaction with sexual encounters. Higher percentage of Ejaculations or Satisfaction in successful sexual intercourse represents better sexual function.
  percentage of successful intercourse
    Successful sexual Intercourse(Ejaculations) | 36 (40) | 54 (45) | 45 (43)
    Successful Sexual Intercourse (Satisfaction) | 22 (34) | 40 (45) | 31 (40)
Male Sexual Health Questionnaire (MSHQ) [Mean (Standard Deviation); unit: units on a scale] — MSHQ, a 25-item questionnaire, assesses sexual function and satisfaction. It consists 5 domains: Erection (3 items, ranging from 0 to 15 (best)), Ejaculation (7 items, ranging from 1 to 35 (best)), Satisfaction (6 items, ranging from 6 to 30 (best)), Sexual desire (4 items, ranging 4-20 (best)), and Sexual activity (3 items, ranging 3-15 (best)). A composite score is the sum of Ejaculation and Satisfaction domains, ranging from 7 to 65 (best), with higher score representing better sexual function and satisfaction.
  units on a scale
    Erection | 6.7 (1.9) | 6.9 (1.8) | 6.8 (1.9)
    Ejaculation | 22.2 (6.6) | 22.2 (7.3) | 22.2 (7.0)
    Sexual satisfaction | 19.5 (5.7) | 18.7 (6.0) | 19.1 (5.8)
    Sexual desire | 8.6 (2.4) | 8.6 (2.5) | 8.6 (2.4)
    Sexual activity | 5.5 (1.4) | 5.6 (1.5) | 5.5 (1.4)
    Composite MSHQ | 41.7 (9.6) | 40.8 (10.6) | 41.2 (10.1)
Quality of Life Specific to Male Erection Difficulties (QOL-MED) [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life for men with Erection Difficulties (QOL-MED) is a cross-cultural instrument to measure quality of life specific to male erection difficulties. The 18 items for this scale were generated from interviews with men with erection difficulties by TH Wagner in 1996. Scores were standardized to 0 to 100. Higher QOL-MED scores reflect better quality of life.
  units on a scale | 47 (25) | 51 (26) | 49 (26)
Marital Interaction scale in CAncer Rehabilitation Evaluation System-Short Form (CARES-SF) [Mean (Standard Deviation); unit: units on a scale] — CAncer Rehabilitation Evaluation System-short form (CARES-SF) marital interaction scale consists of 6 items (range from 0 (best) to 4) and mean of these 6 questions was used to determine intimacy and partner interaction. Lower CARES-SF scores correspond with improved marital interaction.
  units on a scale | 0.91 (0.82) | 0.79 (0.78) | 0.85 (0.80)
Psychological Global Well-Being Index (PGWBI) [Mean (Standard Deviation); unit: units on a scale] — PGWBI consists of 22 items each ranges from 0 (poor) to 5 (good) measuring Quality of Life (QoL). It measures 6 dimensions of perceived well-being and distress: Anxiety (5 questions), Depressed Mood (3 questions), Positive Well-Being (4 questions), Self Control (3 questions), General Health (3 questions), and Vitality (4 questions). An global score is the sum of 6 domains, ranging from 0 (poor QoL) to 110 (good QoL). The PGWBI global score and those of its 6 dimensions are normalized to 0-100. Higher score represents better QoL.
  units on a scale
    Anxiety | 75 (15) | 72 (18) | 74 (17)
    Depressed mood | 86 (14) | 83 (15) | 84 (14)
    Positive well-being | 62 (17) | 61 (19) | 61 (18)
    Self-control | 85 (13) | 84 (14) | 85 (14)
    General health | 73 (16) | 73 (17) | 73 (17)
    Vitality | 65 (15) | 65 (19) | 65 (17)
    Global score | 73 (12) | 72 (14) | 73 (13)
Derogatis Affects Balance Scale (DABS) [Mean (Standard Deviation); unit: units on a scale] — The DABS measures affectivity and affects balance via 4 positive (Joy, Contentment, Vigor, and Affection) and 4 negative (Anxiety, Depression, Guilt, and Hostility) dimensions that reflect basic emotional states. Each domain is scored separately from 0 to 20 with higher scores representing stronger emotional feeling.
  units on a scale
    Joy | 13.0 (3.2) | 12.9 (4.3) | 13.0 (3.8)
    Contentment | 13.1 (2.9) | 12.8 (3.6) | 12.9 (3.2)
    Vigor | 12.2 (3.2) | 12.3 (4.1) | 12.2 (3.7)
    Affection | 14.4 (3.6) | 14.2 (3.8) | 14.3 (3.7)
    Depression | 3.9 (3.3) | 4.7 (3.7) | 4.3 (3.5)
    Anxiety | 5.4 (3.5) | 6.2 (3.1) | 5.8 (3.4)
    Guilt | 4.1 (3.7) | 4.4 (3.9) | 4.3 (3.8)
    Hostiity | 4.5 (3.5) | 4.8 (3.7) | 4.7 (3.6)
Positive Affect Ratio (PAR) in Derogatis Affects Balance Scale (DABS) [Mean (Standard Deviation); unit: ratios] — The DABS measures affectivity and affects balance via 4 positive (Joy, Contentment, Vigor, and Affection) and 4 negative (Anxiety, Depression, Guilt, and Hostility) dimensions that reflect basic emotional states. Positive Affects Ratio (PAR), ranging from 0 to 1, is the proportion of total scores (sum of all 8 domains) that is positive (sum of 4 positive domains). Higher PAR represents better affectivity.
  ratios | 0.75 (0.14) | 0.74 (0.16) | 0.74 (0.15)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Erectile Function Domain Score of the International Index of Erectile Function (IIEF)
Description: IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with Erectile Function domain range of 1 to 30 with higher scores representing better function.
Time Frame: Week 0, week 8, week 11, week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
units on a scale
  Erectile function at week 0: number analyzed (Participants) | 67 | 68
  Erectile function at week 0 | 19.6 (7.2) | 20.1 (7.2)
  Erectile function at week 8: number analyzed (Participants) | 64 | 63
  Erectile function at week 8 | 21.3 (7.4) | 21.3 (8.0)
  Erectile function at week 11: number analyzed (Participants) | 62 | 60
  Erectile function at week 11 | 22.5 (7.0) | 20.1 (8.5)
  Erectile function at week 14: number analyzed (Participants) | 58 | 57
  Erectile function at week 14 | 21.7 (7.9) | 19.8 (8.6)

2. Secondary Outcome: Change From Baseline in Other Domains of International Index of Erectile Function (IIEF)
Description: IIEF is a validated, 15-item questionnaire that assesses 5 domains of sexual function: erectile function (range 1-30), orgasmic function (range 0-10), sexual desire (range 2-10), intercourse satisfaction (range 0-15), and overall sexual satisfaction (range 2-10). Each question was answered on a 6-point or 5-point scale from 0/1 to 5 (best) with a total possible score (sum of 5 domains) range of 5 to 75 with higher scores representing better function.
Time Frame: Week 0, week 8, week 11, week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
units on a scale
  Orgasmic function at week 0 | 7.0 (2.7) | 7.0 (2.6)
  Orgasmic function at week 8: number analyzed (Participants) | 65 | 64
  Orgasmic function at week 8 | 7.6 (2.4) | 7.8 (2.7)
  Orgasmic function at week 11: number analyzed (Participants) | 63 | 62
  Orgasmic function at week 11 | 7.9 (2.5) | 7.4 (3.0)
  Orgasmic function at week 14: number analyzed (Participants) | 60 | 58
  Orgasmic function at week 14 | 7.9 (2.8) | 7.4 (3.1)
  Sexual desire at week 0 | 6.5 (1.9) | 6.7 (1.5)
  Sexual desire at week 8: number analyzed (Participants) | 65 | 64
  Sexual desire at week 8 | 7.0 (1.8) | 7.0 (1.6)
  Sexual desire at week 11: number analyzed (Participants) | 63 | 62
  Sexual desire at week 11 | 7.1 (2.0) | 6.8 (2.0)
  Sexual desire at week 14: number analyzed (Participants) | 60 | 58
  Sexual desire at week 14 | 7.0 (2.0) | 6.8 (2.0)
  Intercourse satisfaction at week 0: number analyzed (Participants) | 69 | 69
  Intercourse satisfaction at week 0 | 9.5 (3.0) | 9.4 (3.4)
  Intercourse satisfaction at week 8: number analyzed (Participants) | 65 | 64
  Intercourse satisfaction at week 8 | 10.1 (3.3) | 9.8 (3.9)
  Intercourse satisfaction at week 11: number analyzed (Participants) | 62 | 62
  Intercourse satisfaction at week 11 | 10.6 (3.3) | 9.5 (4.2)
  Intercourse satisfaction at week 14: number analyzed (Participants) | 60 | 58
  Intercourse satisfaction at week 14 | 10.0 (4.0) | 8.8 (4.2)
  Overall satisfaction at week 0 | 6.4 (2.1) | 6.6 (2.4)
  Overall satisfaction at week 8: number analyzed (Participants) | 64 | 63
  Overall satisfaction at week 8 | 6.8 (2.2) | 7.3 (2.2)
  Overall satisfaction at week 11: number analyzed (Participants) | 63 | 62
  Overall satisfaction at week 11 | 7.4 (2.0) | 7.0 (2.5)
  Overall satisfaction at week 14: number analyzed (Participants) | 60 | 58
  Overall satisfaction at week 14 | 6.7 (2.3) | 7.0 (2.4)
  Composite IIEF at week 0: number analyzed (Participants) | 66 | 68
  Composite IIEF at week 0 | 47 (17) | 50 (18)
  Composite IIEF at week 8: number analyzed (Participants) | 63 | 62
  Composite IIEF at week 8 | 53 (15) | 53 (16)
  Composite IIEF at week 11: number analyzed (Participants) | 62 | 60
  Composite IIEF at week 11 | 56 (14) | 51 (18)
  Composite IIEF at week 14: number analyzed (Participants) | 58 | 57
  Composite IIEF at week 14 | 53 (17) | 50 (18)

3. Secondary Outcome: Change From Baseline in Sexual Encounter Profile (SEP)
Description: Sexual Encounter Profile (SEP) diaries were used to assess frequency of sexual activity, sildenafil use, vaginal penetration, completion of intercourse with ejaculation, and overall satisfaction with sexual encounters. Minimum value is 0 with no maximum limit, wherein higher values representing better sexual encounter.
Time Frame: Week 0, week 8, week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: events/week
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
events/week
  Sexual Encounter Attempts at week 0: number analyzed (Participants) | 62 | 56
  Sexual Encounter Attempts at week 0 | 2.8 (1.5) | 3.0 (1.3)
  Sexual Encounter Attempts at week 8: number analyzed (Participants) | 58 | 53
  Sexual Encounter Attempts at week 8 | 2.8 (1.2) | 3.0 (1.2)
  Sexual Encounter Attempts at week 14: number analyzed (Participants) | 47 | 42
  Sexual Encounter Attempts at week 14 | 3.3 (1.6) | 3.0 (1.2)
  Vaginal Penetration at week 0: number analyzed (Participants) | 62 | 56
  Vaginal Penetration at week 0 | 2.7 (1.4) | 2.6 (0.9)
  Vaginal Penetration at week 8: number analyzed (Participants) | 58 | 53
  Vaginal Penetration at week 8 | 2.4 (1.1) | 2.7 (1.1)
  Vaginal Penetration at week 14: number analyzed (Participants) | 46 | 42
  Vaginal Penetration at week 14 | 2.7 (1.4) | 2.6 (0.9)
  Ejaculation at week 0: number analyzed (Participants) | 62 | 55
  Ejaculation at week 0 | 2.1 (1.6) | 2.2 (1.4)
  Ejaculation at week 8: number analyzed (Participants) | 58 | 53
  Ejaculation at week 8 | 2.3 (1.5) | 2.5 (1.2)
  Ejaculation at week 14: number analyzed (Participants) | 47 | 42
  Ejaculation at week 14 | 2.6 (1.7) | 2.3 (1.3)
  Overall Satisfied with Sexual Encounters at week0: number analyzed (Participants) | 62 | 55
  Overall Satisfied with Sexual Encounters at week0 | 2.0 (1.7) | 1.9 (1.4)
  Overall Satisfied with Sexual Encounters at week8: number analyzed (Participants) | 58 | 53
  Overall Satisfied with Sexual Encounters at week8 | 2.2 (1.5) | 2.3 (1.4)
  Overall Satisfied with Sexual Encounters at wk 14: number analyzed (Participants) | 47 | 41
  Overall Satisfied with Sexual Encounters at wk 14 | 2.8 (1.8) | 2.5 (1.3)

4. Secondary Outcome: Change From Baseline in Successful Sexual Intercourse of Sexual Encounter Profile (SEP)
Description: Sexual Encounter Profile (SEP) diaries were used to assess frequency of sexual activity, sildenafil use, vaginal penetration, completion of intercourse with ejaculation, and overall satisfaction with sexual encounters. Higher percentage of Ejaculations or Satisfaction in successful sexual intercourse represents better sexual function.
Time Frame: Week 0, week 8, week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: percentage of sexual intercourses
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
percentage of sexual intercourses
  Successful Sexual Intercourse (Ejaculations) wk0: number analyzed (Participants) | 62 | 55
  Successful Sexual Intercourse (Ejaculations) wk0 | 76 (37) | 74 (35)
  Successful Sexual Intercourse (Ejaculations) wk8: number analyzed (Participants) | 58 | 53
  Successful Sexual Intercourse (Ejaculations) wk8 | 78 (40) | 84 (29)
  Successful Sexual Intercourse (Ejaculations)wk14: number analyzed (Participants) | 47 | 42
  Successful Sexual Intercourse (Ejaculations)wk14 | 80 (31) | 79 (37)
  Successful Sexual Intercourse (Satisfaction) wk0: number analyzed (Participants) | 62 | 55
  Successful Sexual Intercourse (Satisfaction) wk0 | 69 (39) | 67 (40)
  Successful Sexual Intercourse (Satisfaction) wk8: number analyzed (Participants) | 58 | 53
  Successful Sexual Intercourse (Satisfaction) wk8 | 76 (39) | 75 (35)
  Successful Sexual Intercourse (Satisfaction)wk14: number analyzed (Participants) | 47 | 41
  Successful Sexual Intercourse (Satisfaction)wk14 | 83 (34) | 83 (33)

5. Secondary Outcome: Change From Baseline in Men's Sexual Health Questionnaire (MSHQ)
Description: MSHQ, a 25-item questionnaire, assesses sexual function and satisfaction. It consists 5 domains: Erection (3 items, ranging from 0 to 15 (best)), Ejaculation (7 items, ranging from 1 to 35 (best)), Satisfaction (6 items, ranging from 6 to 30 (best)), Sexual desire (4 items, ranging 4-20 (best)), and Sexual activity (3 items, ranging 3-15 (best)). A composite score is the sum of Ejaculation and Satisfaction domains, ranging from 7 to 65 (best), with higher score representing better sexual function and satisfaction.
Time Frame: Week 0, Week 8, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
units on a scale
  Erectile at week 0: number analyzed (Participants) | 61 | 58
  Erectile at week 0 | 5.3 (3.4) | 5.9 (2.9)
  Erectile at week 8: number analyzed (Participants) | 57 | 50
  Erectile at week 8 | 6.3 (3.8) | 6.9 (3.7)
  Erectile at week 14: number analyzed (Participants) | 52 | 49
  Erectile at week 14 | 6.9 (3.2) | 7.2 (3.6)
  Ejaculation at week 0: number analyzed (Participants) | 69 | 69
  Ejaculation at week 0 | 26.8 (5.7) | 26.1 (7.1)
  Ejaculation at week 8: number analyzed (Participants) | 64 | 62
  Ejaculation at week 8 | 28.3 (4.6) | 27.8 (5.9)
  Ejaculation at week 14: number analyzed (Participants) | 60 | 58
  Ejaculation at week 14 | 28.4 (5.4) | 26.9 (6.2)
  Sexual satisfaction at week 0: number analyzed (Participants) | 69 | 69
  Sexual satisfaction at week 0 | 22.1 (5.2) | 21.6 (6.2)
  Sexual satisfaction at week 8: number analyzed (Participants) | 64 | 64
  Sexual satisfaction at week 8 | 22.3 (5.2) | 22.4 (5.9)
  Sexual satisfaction at week 14: number analyzed (Participants) | 59 | 56
  Sexual satisfaction at week 14 | 22.5 (6.3) | 21.5 (6.2)
  Sexual desire at week 0: number analyzed (Participants) | 68 | 70
  Sexual desire at week 0 | 9.9 (2.4) | 10.3 (2.8)
  Sexual desire at week 8: number analyzed (Participants) | 65 | 64
  Sexual desire at week 8 | 10.5 (2.2) | 10.7 (2.5)
  Sexual desire at week 14: number analyzed (Participants) | 60 | 57
  Sexual desire at week 14 | 10.5 (2.6) | 10.1 (2.7)
  Sexual activity at week 0 | 7.0 (1.5) | 6.7 (1.7)
  Sexual activity at week 8: number analyzed (Participants) | 64 | 64
  Sexual activity at week 8 | 7.1 (1.4) | 6.9 (1.6)
  Sexual activity at week 14: number analyzed (Participants) | 60 | 58
  Sexual activity at week 14 | 7.0 (1.6) | 6.5 (1.8)
  Composite MSHQ at week 0: number analyzed (Participants) | 68 | 68
  Composite MSHQ at week 0 | 48.8 (9.1) | 47.7 (11.4)
  Composite MSHQ at week 8: number analyzed (Participants) | 63 | 62
  Composite MSHQ at week 8 | 50.6 (7.8) | 50.2 (9.5)
  Composite MSHQ at week 14: number analyzed (Participants) | 59 | 56
  Composite MSHQ at week 14 | 51.1 (9.4) | 48.5 (10.5)

6. Secondary Outcome: Change From Baseline in Quality of Life Specific to Male Erection Difficulties (QOL-MED)
Description: The Quality of Life for men with Erection Difficulties (QOL-MED) is a cross-cultural instrument to measure quality of life specific to male erection difficulties. The 18 items for this scale were generated from interviews with men with erection difficulties by TH Wagner in 1996. Higher QOL-MED scores reflect better quality of life. Scores were standardized to range of 0 to 100.
Time Frame: Week 0, Week 8, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
units on a scale
  QOL-MED scale at week 0: number analyzed (Participants) | 69 | 70
  QOL-MED scale at week 0 | 56 (26) | 62 (26)
  QOL-MED scale at week 8: number analyzed (Participants) | 65 | 62
  QOL-MED scale at week 8 | 65 (25) | 70 (26)
  QOL-MED scale at week 14: number analyzed (Participants) | 58 | 58
  QOL-MED scale at week 14 | 66 (25) | 69 (25)

7. Secondary Outcome: Change From Baseline in Marital Interaction Scale of CAncer Rehabilitation Evaluation System-Short Form (CARES-SF)
Description: CAncer Rehabilitation Evaluation System-short form (CARES-SF) marital interaction scale consists of 6 items (range from 0 (best) to 4) and mean of these 6 questions was used to determine intimacy and partner interaction. Lower CARES-SF scores correspond with improved marital interaction.
Time Frame: Week 0, Week 8, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
units on a scale
  CARES-SF: Marital relationship at week 0: number analyzed (Participants) | 69 | 70
  CARES-SF: Marital relationship at week 0 | 0.79 (0.70) | 0.74 (0.77)
  CARES-SF: Marital relationship at week 8: number analyzed (Participants) | 64 | 63
  CARES-SF: Marital relationship at week 8 | 0.86 (0.74) | 0.79 (0.95)
  CARES-SF: Marital relationship at week 14: number analyzed (Participants) | 59 | 58
  CARES-SF: Marital relationship at week 14 | 0.81 (0.81) | 0.79 (0.79)

8. Secondary Outcome: Change From Baseline in Psychological General Well-Being Index Score (PGWBI)
Description: Well-being and mood were assessed using the Psychological General Well-Being Index (PGWBI), a 22-item questionnaire that evaluated six dimensions of self-reported wellness: Anxiety (5 questions), Depressed Mood (3 questions), Positive Well-Being (4 questions), Self Control (3 questions), General Health (3 questions), and Vitality (4 questions). Higher scores in each dimension reflect increasing well-being. A global score (ranging from 0 (poor QoL) to 110 (good QoL)) was calculated as the sum of each domain score. The global score and those of its 6 dimensions were normalized to a 100% scale to facilitate comparison.
Time Frame: Week 0, Week 8, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
units on a scale
  Positive Well-being at week 0: number analyzed (Participants) | 70 | 69
  Positive Well-being at week 0 | 60 (19) | 63 (18)
  Positive Well-being at week 8: number analyzed (Participants) | 65 | 62
  Positive Well-being at week 8 | 65 (18) | 63 (18)
  Positive Well-being at week 14: number analyzed (Participants) | 60 | 58
  Positive Well-being at week 14 | 64 (20) | 60 (21)
  Depressed Mood at week 0: number analyzed (Participants) | 70 | 68
  Depressed Mood at week 0 | 86 (16) | 86 (15)
  Depressed Mood at week 8: number analyzed (Participants) | 65 | 63
  Depressed Mood at week 8 | 85 (15) | 86 (18)
  Depressed Mood at week 14: number analyzed (Participants) | 60 | 58
  Depressed Mood at week 14 | 85 (18) | 83 (18)
  General Health at week 0: number analyzed (Participants) | 70 | 69
  General Health at week 0 | 72 (16) | 74 (17)
  General Health at week 8: number analyzed (Participants) | 65 | 62
  General Health at week 8 | 73 (19) | 75 (18)
  General Health at week 14: number analyzed (Participants) | 60 | 58
  General Health at week 14 | 72 (17) | 70 (23)
  Anxiety at week 0 | 76 (15) | 76 (19)
  Anxiety at week 8: number analyzed (Participants) | 65 | 63
  Anxiety at week 8 | 76 (15) | 76 (20)
  Anxiety at week 14: number analyzed (Participants) | 60 | 58
  Anxiety at week 14 | 77 (15) | 72 (22)
  Self Control at week 0: number analyzed (Participants) | 70 | 69
  Self Control at week 0 | 86 (14) | 84 (15)
  Self Control at week 8: number analyzed (Participants) | 65 | 63
  Self Control at week 8 | 86 (17) | 86 (15)
  Self Control at week 14: number analyzed (Participants) | 60 | 58
  Self Control at week 14 | 87 (15) | 84 (16)
  Vitality at week 0: number analyzed (Participants) | 70 | 68
  Vitality at week 0 | 66 (17) | 68 (18)
  Vitality at week 8: number analyzed (Participants) | 65 | 63
  Vitality at week 8 | 68 (17) | 69 (17)
  Vitality at week 14: number analyzed (Participants) | 60 | 58
  Vitality at week 14 | 69 (19) | 67 (19)
  Global Score at week 0: number analyzed (Participants) | 70 | 67
  Global Score at week 0 | 73 (13) | 74 (15)
  Global Score at week 8: number analyzed (Participants) | 65 | 61
  Global Score at week 8 | 75 (14) | 75 (14)
  Global Score at week 14: number analyzed (Participants) | 60 | 58
  Global Score at week 14 | 75 (14) | 72 (17)

9. Secondary Outcome: Change From Baseline in Derogatis Affects Balance Scale (DABS)
Description: The Derogatis Affects Balance Scale (DABS) is a 40-item mood inventory and consists of 4 positive affect dimensions (joy, contentment, vigor, and affection) as well as 4 negative affect dimensions(anxiety, depression, guilt, and hostility). Each domain was calculated as the sum of 5-items and could range from 0 to 20, wherein higher scores indicate greater affectivity.
Time Frame: Week 0, Week 8, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
units on a scale
  Joy at week 0: number analyzed (Participants) | 67 | 69
  Joy at week 0 | 12.7 (3.3) | 13.1 (3.4)
  Joy at week 8: number analyzed (Participants) | 65 | 62
  Joy at week 8 | 13.1 (3.1) | 13.5 (3.7)
  Joy at week 14: number analyzed (Participants) | 58 | 54
  Joy at week 14 | 13.2 (3.2) | 12.7 (3.9)
  Contentment at week 0: number analyzed (Participants) | 68 | 69
  Contentment at week 0 | 12.8 (3.2) | 13.2 (3.3)
  Contentment at week 8: number analyzed (Participants) | 63 | 64
  Contentment at week 8 | 13.4 (2.8) | 13.7 (3.5)
  Contentment at week 14: number analyzed (Participants) | 59 | 54
  Contentment at week 14 | 13.3 (3.2) | 12.8 (4.2)
  Vigor at week 0: number analyzed (Participants) | 68 | 68
  Vigor at week 0 | 11.8 (3.3) | 12.0 (3.6)
  Vigor at week 8: number analyzed (Participants) | 65 | 64
  Vigor at week 8 | 12.5 (3.1) | 13.0 (3.8)
  Vigor at week 14: number analyzed (Participants) | 59 | 56
  Vigor at week 14 | 12.6 (3.6) | 12.6 (4.1)
  Affection at week 0: number analyzed (Participants) | 68 | 69
  Affection at week 0 | 13.9 (3.3) | 14.6 (3.4)
  Affection at week 8: number analyzed (Participants) | 64 | 62
  Affection at week 8 | 14.2 (3.4) | 14.7 (3.8)
  Affection at week 14: number analyzed (Participants) | 57 | 54
  Affection at week 14 | 14.2 (3.9) | 14.5 (3.7)
  Depression at week 0 | 4.1 (3.9) | 3.9 (3.7)
  Depression at week 8: number analyzed (Participants) | 65 | 63
  Depression at week 8 | 4.1 (3.5) | 4.3 (4.2)
  Depression at week 14: number analyzed (Participants) | 59 | 55
  Depression at week 14 | 4.2 (4.0) | 4.1 (3.8)
  Anxiety at week 0: number analyzed (Participants) | 69 | 68
  Anxiety at week 0 | 4.9 (3.3) | 5.5 (3.8)
  Anxiety at week 8: number analyzed (Participants) | 65 | 63
  Anxiety at week 8 | 5.1 (3.4) | 5.6 (3.7)
  Anxiety at week 14: number analyzed (Participants) | 59 | 56
  Anxiety at week 14 | 4.9 (3.5) | 5.8 (3.8)
  Guilt at week 0: number analyzed (Participants) | 68 | 67
  Guilt at week 0 | 3.4 (3.6) | 4.1 (3.9)
  Guilt at week 8: number analyzed (Participants) | 64 | 62
  Guilt at week 8 | 3.7 (3.6) | 4.5 (4.4)
  Guilt at week 14: number analyzed (Participants) | 58 | 55
  Guilt at week 14 | 3.8 (4.1) | 3.7 (3.8)
  Hostility at week 0: number analyzed (Participants) | 67 | 68
  Hostility at week 0 | 4.7 (3.4) | 4.3 (3.7)
  Hostility at week 8: number analyzed (Participants) | 63 | 61
  Hostility at week 8 | 4.6 (3.3) | 4.6 (4.3)
  Hostility at week 14: number analyzed (Participants) | 59 | 56
  Hostility at week 14 | 4.7 (3.9) | 4.4 (3.8)

10. Secondary Outcome: Change From Baseline in Positive Affects Ratio (PAR) of Derogatis Affects Balance Scale (DABS)
Description: The Derogatis Affects Balance Scale (DABS) is a 40-item mood inventory and consists of 4 positive affect dimensions (joy, contentment, vigor, and affection) as well as 4 negative affect dimensions(anxiety, depression, guilt, and hostility). Positive Affects Ratio (PAR), ranging from 0 to 1, is the proportion of total scores (sum of all 8 domains) that is positive (sum of 4 positive domains). Higher PAR represents better affectivity.
Time Frame: Week 0, Week 8, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: ratios
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
ratios
  Positive Affect Ratio at week 0: number analyzed (Participants) | 61 | 65
  Positive Affect Ratio at week 0 | 0.75 (0.15) | 0.76 (0.16)
  Positive Affect Ratio at week 8: number analyzed (Participants) | 60 | 58
  Positive Affect Ratio at week 8 | 0.76 (0.16) | 0.77 (0.17)
  Positive Affect Ratio at week 14: number analyzed (Participants) | 55 | 47
  Positive Affect Ratio at week 14 | 0.78 (0.17) | 0.76 (0.18)

11. Other Pre Specified Outcome: Change From Baseline in Total Testosterone
Description: Total testosterone levels were measured between 7:30 and 10:10 a.m. using a liquid chromatography-tandem mass spectrometry assay certified by the Centers for Disease Control and Prevention's Hormone Standardization Program.
Time Frame: Week 0, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
ng/dL
  Total Testosterone at week 0: number analyzed (Participants) | 64 | 61
  Total Testosterone at week 0 | 364 (192) | 347 (141)
  Total Testosterone at week 14: number analyzed (Participants) | 58 | 57
  Total Testosterone at week 14 | 649 (411) | 339 (155)

12. Other Pre Specified Outcome: Change From Baseline in Free Testosterone
Description: Free testosterone levels were calculated from total testosterone at screening and equilibrium dialysis at randomization and at trial end.
Time Frame: Week 0, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
pg/mL
  Free Testosterone at week 0: number analyzed (Participants) | 64 | 61
  Free Testosterone at week 0 | 110 (79) | 101 (36)
  Free Testosterone at week 14: number analyzed (Participants) | 58 | 57
  Free Testosterone at week 14 | 239 (197) | 103 (63)

13. Other Pre Specified Outcome: Change From Baseline in Sex Hormone Binding Globulin (SHBG)
Time Frame: Week 0, Week 14
Population: All available data expressed as absolute value at the given time-point.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 70 | 70
nmol/L
  SHBG at week 0: number analyzed (Participants) | 64 | 61
  SHBG at week 0 | 32.2 (14.7) | 27.5 (14.6)
  SHBG at week 14: number analyzed (Participants) | 58 | 57
  SHBG at week 14 | 32 (16) | 28 (15)

ADVERSE EVENTS:
Arm/Group | Testosterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 2/70 | 4/70
Other Adverse Events (participants affected / at risk) | 27/70 | 13/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone (N=70) | Placebo (N=70)
Chest pain (Cardiac disorders) | 1 | 0
Acute cholecystitis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Incisional hernia repair (Surgical and medical procedures) | 0 | 1
Fever (General disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Chills (Musculoskeletal and connective tissue disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone (N=70) | Placebo (N=70)
Upper respiratory tract infection (Infections and infestations) | 10 | 7
Keen pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Tooth ache (Gastrointestinal disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No